CLINICAL TRIAL: NCT00508235
Title: Quality of Friendships in Children With Neurofibromatosis: Relationship to Disease Severity
Brief Title: Quality of Friendships in Children With Neurofibromatosis
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0791
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Neurofibromatosis
Keywords: Neurofibromatosis; Quality of Friendships; Disease Severity; Questionnaire; NF-1
MeSH Terms: conditions — Neurofibromatoses | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Quality of Friendships: Patients with Neurofibromatosis, type 1 (NF-1) between the ages of 8 and 18 years old.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire about the patient's relationship with their best friend.
  Other Names: Survey

SUMMARY:
The aim of this study is to determine if children with a higher disease severity have lower quality friendships than children who are less severely affected and children who are unaffected. Researchers will test the hypothesis that the quality of friendships is inversely related to their disease severity.

Specific Aims:

1. To use the FQQ to determine if the quality of friendships in children with NF1 is lower than the quality of friendships in unaffected children.
2. To use a disease severity scale and the FQQ to determine if children who are less severely affected have higher friendship qualities than children who are more severely affected.

DETAILED DESCRIPTION:
You (your) child will be asked to complete a short questionnaire (40 questions) about their relationship with their best friend. Doctors will review your (child's) medical chart to find out how severe the disease is, so that this may be compared to the answers you have (your child has) given on the friendship questionnaire.

This is an Investigational Study. About 90-100 children and adolescents with NF-1 will be asked to take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1) Patients with a clinical diagnosis of neurofibromatosis, type 1 (NF-1) who are between the ages of 8 and 18 years will be eligible. Patients must be English or Spanish speaking (test instrument will be translated into Spanish), and be able to read.

Exclusion Criteria:

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study participants with Neurofibromatosis, type 1 (NF-1) between the ages of 8 and 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2004-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Disease severity scale and Friendship Quality Questionnaire (FQQ) | Questionnaire completion by patient and chart review by doctor for disease severity scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Bartlett D. Moore, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org